CLINICAL TRIAL: NCT01870297
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of LY3025876 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3025876 in Participants With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14347; I6D-MC-SMRB (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-31; First posted 2013-06-06 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY3025876 (Experimental): Part A: 0.5 milligram (mg), 1.5 mg, 5 mg, and 15 mg of LY3025876 administered as once daily (QD) subcutaneous (SQ) injections for up to 28 days.
  Interventions: Drug: LY3025876
- Placebo (Placebo Comparator): Part B: Placebo matching LY3025876 administered as QD SQ injections for up to 28 days
  Interventions: Drug: Placebo
- LY3025876 + Liraglutide (Experimental): Part B: 5.0 mg of LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
  Interventions: Drug: LY3025876; Drug: Liraglutide
- Placebo + Liraglutide (Placebo Comparator): Part B: Placebo doses matching LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
  Interventions: Drug: Placebo; Drug: Liraglutide

INTERVENTIONS:
Drug: LY3025876 — Administered SQ
  Arms: LY3025876; LY3025876 + Liraglutide
Drug: Placebo — Administered SQ
  Arms: Placebo; Placebo + Liraglutide
Drug: Liraglutide — Administered SQ
  Arms: LY3025876 + Liraglutide; Placebo + Liraglutide

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY3025876 given alone (Part A) and in combination with liraglutide (Part B) in participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study will also evaluate how much of the study drug enters the blood stream and how long it takes for the body to remove the study drug. Information about any side effects that may occur will also be collected. Participants will continue their usual diet and exercise program and may remain on their physician-prescribed dose of metformin.

Each part of the study is expected to last 10 to 12 weeks on average, not including screening. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (T2DM) as determined by the investigator, controlled with diet or exercise alone or on a stable dose of metformin for at least 30 days
* Have a body mass index (BMI) greater than or equal to 23 and less than or equal to 45 kilograms per square meter (kg/m^2) at screening
* Have a supine blood pressure reading at screening of between 90-160 millimeter of mercury (mmHg) (systolic) and 40-95 mmHg (diastolic)
* Women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause

Exclusion Criteria:

* Have taken LY3025876 or investigational drugs like it (for example, other fibroblast growth factor-21 [FGF21]-related drugs) or have known allergies to these drugs
* History or presence of bone disease (including osteoporosis or unhealed fractures)
* Current active treatment of periodontal disease
* Have had a significant change in weight, defined as a gain or loss of at least 4 kilogram (kg) (9 pounds) in the last 3 months
* Have had greater than 1 episode of severe hypoglycemia within 6 months of screening that required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions or had a seizure or coma
* Have known allergies or a history of intolerance to liraglutide, glucagon-like peptide 1 (GLP-1) analogues, or other related compounds
* Have a history of acute or chronic pancreatitis
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dose escalation was planned for 20 milligrams (mg) of LY3025876 but dose escalation was only up to 15 mg LY3025876.
Groups:
- Placebo Part A: Part A Placebo for LY3025876 administered as once daily (QD) subcutaneous (SQ) injections for up to 28 days.
- 0.5 mg LY3025876: Part A: 0.5 mg of LY3025876 administered as QD SQ injections for up to 28 days.
- 1.5 mg LY3025876: Part A: 1.5 mg of LY3025876 administered as QD SQ injections for up to 28 days.
- 5.0 mg LY3025876: Part A: 5.0 mg of LY3025876 administered as QD SQ injections for up to 28 days.
- 15 mg LY3025876: Part A: 15 mg of LY3025876 administered as QD SQ injections for up to 28 days.
- 5.0 mg LY3025876 + Lirgalutide: Part B: 5.0 mg LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
Period: Overall Study
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo + Liraglutide | 5.0 mg LY3025876 + Lirgalutide
Started | 11 | 15 | 8 | 9 | 10 | 9 | 10
Completed | 11 | 8 | 7 | 9 | 7 | 8 | 8
Not Completed | 0 | 7 | 1 | 0 | 3 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Sponsor Decision | 0 | 6 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Part A: Part A Placebo for LY3025876 administered as QD SQ injections for up to 28 days.
- 5.0 mg LY3025876 + Liraglutide: Part B:5.0 mg LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo + Liraglutide | 5.0 mg LY3025876 + Liraglutide | Total
Number analyzed (Participants) | 11 | 15 | 8 | 9 | 10 | 9 | 10 | 72
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age Part A | 53.4 (9.6) | 55.8 (7.6) | 53.3 (7.2) | 61.9 (5.5) | 55.3 (6.8) | NA (NA) — see Part B category | NA (NA) — see Part B category | 55.8 (7.8)
  Age Part B | NA (NA) — see Part A category | NA (NA) — see Part A category | NA (NA) — see Part A category | NA (NA) — see Part A category | NA (NA) — see Part A category | 53.2 (8.9) | 54.4 (5.5) | 53.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 2 | 2 | 2 | 3 | 22
  Male | 7 | 10 | 4 | 7 | 8 | 7 | 7 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 7 | 6 | 6 | 6 | 3 | 51
  Not Hispanic or Latino | 1 | 2 | 1 | 3 | 4 | 3 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 0 | 1 | 4 | 8
  White | 11 | 13 | 8 | 7 | 10 | 8 | 5 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 15 | 8 | 9 | 10 | 9 | 10 | 72
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent of HbA1c]
  HbA1c Part A | 8.64 (0.65) | 8.39 (0.93) | 8.43 (0.88) | 8.94 (1.19) | 8.67 (0.92) | NA (NA) — see Part B category | NA (NA) — see Part B category | 8.59 (0.91)
  HbA1c Part B | NA (NA) — see part A category | NA (NA) — see part A category | NA (NA) — see part A category | NA (NA) — see part A category | NA (NA) — see part A category | 8.56 (0.77) | 8.05 (0.86) | 8.29 (0.84)
Fasting Serum Glucose (FSG) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)]
  FSG Part A | 164.43 (31.59) | 148.08 (19.14) | 181.27 (47.84) | 175.74 (75.99) | 145.66 (23.22) | NA (NA) — see part B below | NA (NA) — see part B below | 161.63 (42.87)
  FSG Part B | NA (NA) — see Part A above | NA (NA) — see Part A above | NA (NA) — see Part A above | NA (NA) — see Part A above | NA (NA) — see Part A above | 159.73 (36.54) | 152.22 (26.62) | 155.78 (31.02)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Predose on Day 1 up to Day 56 in each Part
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo Part A: Part A: Placebo for LY3025876 administered as QD SQ injections for up to 28 days.
- 5.0 mg LY3025876 + Liraglutide: Part B: 5.0 mg LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo + Liraglutide | 5.0 mg LY3025876 + Liraglutide
Number analyzed (Participants) | 11 | 15 | 8 | 9 | 10 | 9 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time 0 to 24 Hours (AUC[0-24]) of LY3025876
Description: AUC(0-24) of individual participants was calculated by equation Area Under Concentration (AUC)=Dose/CL, where the clearance (CL) was estimated using a population PK model.
Time Frame: Predose and 0.5 hour(hr), 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, and 24 hr Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable AUC 0-24 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Groups:
- LY3025876 + Liraglutide: Part B: 5.0 mg LY3025876 and 1.8 mg liraglutide administered as separate QD SQ injections for up to 28 days, after titration of liraglutide over 2 weeks.
Arm/Group | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | LY3025876 + Liraglutide
Number analyzed (Participants) | 15 | 8 | 9 | 8 | 10
nanograms*hour/milliliter (ng*hr/mL) | 51.5 (61.1) | 207 (51.2) | 622 (42.3) | 1930 (32.4) | 525 (37.8)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3025876
Time Frame: Days 1 and 28: Predose and 0.5 hr, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, and 24 hr Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable Cmax PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | 5.0 mg LY3025876 + Liraglutide
Number analyzed (Participants) | 14 | 8 | 9 | 10 | 9
nanogram/milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 13 | 8 | 9 | 9 | 8
  Day 1 | 3.90 (33.7) | 17.5 (43.7) | 45.1 (39.2) | 126 (44.3) | 40.3 (48.3)
  Day 28: number analyzed (Participants) | 7 | 8 | 9 | 5 | 9
  Day 28 | 4.87 (85.7) | 14.2 (46.1) | 51.9 (31.3) | 185 (26.8) | 44.8 (53.8)

4. Secondary Outcome: Part A and Part B: Immunogenicity: The Number of Participants With Anti-LY3025876 Antibodies
Time Frame: Predose on Day 7, 14, 28, 56, and 180
Population: All randomized participants who received at least one dose of study drug in Part A and Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo + Liraglutide | 5.0 mg LY3025876 + Liraglutide
Number analyzed (Participants) | 11 | 15 | 8 | 9 | 10 | 9 | 10
Participants
  Positive Antibodies Day 7 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Positive Antibodies Day 14 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Positive Antibodies Day 28 | 0 | 1 | 2 | 2 | 6 | 0 | 1
  Positive Antibodies Day 56 | 0 | 1 | 4 | 2 | 6 | 0 | 1
  Positive Antibodies Day 180 | 0 | 0 | 0 | 1 | 4 | 0 | 0

5. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline to Day 28 in Fasting Glucose
Description: Least Squares Mean (LS) Mean change from baseline in fasting glucose was modeled using Mixed Effect Model Repeat Measurement (MMRM) analysis with fixed effects of baseline, treatment, day, treatment*day interaction, and participant as a random effect.
Time Frame: Baseline, Day 28
Population: All randomized participants who received one dose of study drug and had evaluable PD data baseline and at least 1 post-baseline data in fasting glucose.
Measure: Least Squares Mean (Standard Error); unit: milligram/deciliter (mg/dL)
Groups:
- Placebo Part B: Part B: Placebo matching LY3025876 administered as QD SQ injections for up to 28 days
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo Part B | 5.0 mg LY3025876 + Liraglutide
Number analyzed (Participants) | 11 | 7 | 8 | 9 | 6 | 8 | 9
milligram/deciliter (mg/dL) | 3.52 (8.41) | 18.08 (10.02) | 0.12 (9.92) | -14.50 (9.33) | 22.96 (11.51) | 11.72 (5.94) | 6.32 (5.64)

ADVERSE EVENTS:
Arm/Group | Placebo Part A | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5.0 mg LY3025876 | 15 mg LY3025876 | Placebo Part B | Placebo + Liraglutide
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/8 | 0/9 | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/11 | 7/15 | 8/8 | 9/9 | 10/10 | 9/9 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Part A (N=11) | 0.5 mg LY3025876 (N=15) | 1.5 mg LY3025876 (N=8) | 5.0 mg LY3025876 (N=9) | 15 mg LY3025876 (N=10) | Placebo Part B (N=9) | Placebo + Liraglutide (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 9 (10) | 0 (0) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (14) | 2 (3) | 2 (8)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (2)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 1 (2) | 1 (5)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food aversion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days